CLINICAL TRIAL: NCT04440163
Title: A PHASE 3, RANDOMIZED, ACTIVE-CONTROLLED, OBSERVER-BLINDED TRIAL TO ASSESS THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MenABCWY IN HEALTHY PARTICIPANTS ≥10 TO <26 YEARS OF AGE
Brief Title: MenABCWY Noninferiority Study in Healthy Participants ≥10 to <26 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3511001; 2019-004313-13 (EudraCT Number)
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Meningococcal Vaccine
MeSH Terms: interventions — Sodium Chloride; MenB-FHbp vaccine; MenACWY-CRM vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 1-Immuno Subset (ACWY Naive,MenABCWY/Saline) (Experimental): ACWY Naive subjects, MenABCWY/Saline
  Interventions: Biological: MenABCWY; Biological: Saline
- 2-Immuno Subset (ACWY Naive, Trumenba/MenACWY-CRM) (Experimental): ACWY Naive subjects, Trumenba/MenACWY-CRM
  Interventions: Biological: Trumenba; Biological: MenACWY-CRM
- 3-Immuno Subset (ACWY Experienced,MenABCWY/Saline) (Experimental): ACWY Experienced subjects, MenABCWY/Saline
  Interventions: Biological: MenABCWY; Biological: Saline
- 4-Immuno Subset (ACWY Experienced,Trumenba/MenACWY-CRM) (Experimental): ACWY Experienced subjects, Trumenba/MenACWY-CRM
  Interventions: Biological: Trumenba; Biological: MenACWY-CRM
- 5-Safety Subset (ACWY Naive,MenABCWY/Saline) (Experimental): ACWY Naive subjects, MenABCWY/Saline
  Interventions: Biological: MenABCWY; Biological: Saline
- 6-Safety Subset (ACWY Naive,Trumenba/MenACWY-CRM) (Experimental): ACWY Naive subjects, Trumenba/MenACWY-CRM
  Interventions: Biological: Trumenba; Biological: MenACWY-CRM
- 7-Safety Subset (ACWY Experienced,MenABCWY/Saline) (Experimental): ACWY Experienced subjects, MenABCWY/Saline
  Interventions: Biological: MenABCWY; Biological: Saline
- 8-Safety Subset (ACWY Experienced,Trumenba/MenACWY-CRM) (Experimental): ACWY Experienced subjects, Trumenba/MenACWY-CRM
  Interventions: Biological: Trumenba; Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenABCWY — N meningitidis groups A, B, C, W, and Y vaccine
  Arms: 1-Immuno Subset (ACWY Naive,MenABCWY/Saline); 3-Immuno Subset (ACWY Experienced,MenABCWY/Saline); 5-Safety Subset (ACWY Naive,MenABCWY/Saline); 7-Safety Subset (ACWY Experienced,MenABCWY/Saline)
Biological: Saline — Placebo
  Arms: 1-Immuno Subset (ACWY Naive,MenABCWY/Saline); 3-Immuno Subset (ACWY Experienced,MenABCWY/Saline); 5-Safety Subset (ACWY Naive,MenABCWY/Saline); 7-Safety Subset (ACWY Experienced,MenABCWY/Saline)
Biological: Trumenba — Bivalent recombinant lipoprotein 2086 vaccine
  Arms: 2-Immuno Subset (ACWY Naive, Trumenba/MenACWY-CRM); 4-Immuno Subset (ACWY Experienced,Trumenba/MenACWY-CRM); 6-Safety Subset (ACWY Naive,Trumenba/MenACWY-CRM); 8-Safety Subset (ACWY Experienced,Trumenba/MenACWY-CRM)
Biological: MenACWY-CRM — Meningococcal group A, C, W-135, and Y conjugate vaccine
  Arms: 2-Immuno Subset (ACWY Naive, Trumenba/MenACWY-CRM); 4-Immuno Subset (ACWY Experienced,Trumenba/MenACWY-CRM); 6-Safety Subset (ACWY Naive,Trumenba/MenACWY-CRM); 8-Safety Subset (ACWY Experienced,Trumenba/MenACWY-CRM)

SUMMARY:
The aim of this study is to determine the immunologic noninferiority of MenABCWY to licensed vaccines Trumenba and MenACWY-CRM (Menveo) by assessing the safety and immunogenicity of MenABCWY and the comparators in both ACWY-naïve and ACWY-experienced healthy participants ≥10 to <26 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged >=10 and <26 years at the time of randomization.
* Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
* Negative urine pregnancy test for all female subjects.
* ACWY-naïve participants: Participants who have never received a prior dose of a meningococcal vaccine containing ACWY serogroups.
* ACWY-experienced participants: Participants who have received not more than 1 prior dose, no sooner than 4 years prior to the date of randomization of Menactra or Menveo.

Exclusion Criteria:

* Previous vaccination with any meningococcal group B vaccine, any purely polysaccharide (nonconjugate) meningococcal vaccine, or monovalent/bivalent meningococcal vaccine.- Subjects receiving any allergen immunotherapy with a non-licensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
* A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects in the United States with terminal complement deficiency are excluded from participation in this study.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Current chronic use of systemic antibiotics.
* Participation in other studies involving investigational drug(s) or investigational vaccine(s) within 28 days prior to study entry and/or during study participation.
* Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
* History of microbiologically proven disease caused by N meningitidis or Neisseria gonorrhoeae.
* Receipt of any blood products, including immunoglobulin, within 6 months before the first study vaccination.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2431 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (77):
- United States (60):
  - Alabama Clinical Therapeutics, LLC, Birmington Pediatric Assocaites, Birmingham, Alabama
  - Central Research Associates, Inc., Birmingham, Alabama
  - Fiel Family and Sports Medicine, PC/CCT Research, Tempe, Arizona
  - Velocity Clinical Research (Banning), Banning, California
  - Madera Family Medical Group, Madera, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Center for Clinical Trials, Paramount, California
  - Optumcare Colorado Springs, LLC, Colorado Springs, Colorado
  - ALL Medical Research, LLC, Cooper City, Florida
  - Alliance for MultiSpecialty Research, LLC - Miami, Coral Gables, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Altus Research, Lake Worth, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Healthy Life Research, Inc., Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Crystal Biomedical Research, LLC, Miami Lakes, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - PAS Research, Tampa, Florida
  - Tekton Research, Inc., Chamblee, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Saltzer Health, Nampa, Idaho
  - MOC Research, Mishawaka, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - The Iowa Clinic, Ankeny, Iowa
  - The Iowa Clinic, West Des Moines, Iowa
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Michael W. Simon, MD, PSC, Lexington, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Acorn to Oak Pediatrics - ACC Pediatric Research, Haughton, Louisiana
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Skyline Medical Center, PC/CCT Research, Elkhorn, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Binghamton, New York
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Liberty Family Practice, Erie, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Accellacare US Inc., Mt. Pleasant, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Family Medicine Associates of Texas, Carrollton, Texas
  - AIM Trials, LLC, Plano, Texas
  - North Texas Family Medicine, Plano, Texas
  - Tekton Research, San Antonio, Texas
  - Olympus Family Medicine/CCT Research, Holladay, Utah
  - Pediatric Care, Provo, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
- Czechia (6):
  - SANARE s.r.o, České Budějovice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - MUDr. Katerina Stichhauerova s.r.o., Pardubice
  - Medicentrum 6 s.r.o., Prague
  - Praktik Pb s.r.o., Příbram
- Aarhus Universitetshospital, Aarhus N, Denmark
- Hungary (5):
  - DRC Gyógyszervizsgáló Központ Kft., Balatonfüred
  - ClinTrial Audit Kft., Klinikai Farmakologiai Intezet, Vedooltasi Ambulancia, Debrecen
  - Coronella Orvosi Centrum / Trial Pharma Kft., Gyula
  - CRU Hungary Kft., Miskolc
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
- Poland (5):
  - Centrum Badan Klinicznych JCI, Krakow
  - Przylądek Zdrowia, Krakow
  - Niepubliczny Zaklad Lecznictwa Ambulatoryjnego MICHALKOWICE, Siemianowice Śląskie
  - Szpital im. Sw. Jadwigi Slaskiej w Trzebnicy, Trzebnica
  - Niepubliczny Zaklad Opieki Zdrowotnej "Salmed", Łęczna

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3511001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2431 participants were enrolled and randomized in the study of which 18 participants did not receive any vaccination. Out of 2431 participants, 2413 participants received at least 1 dose of vaccination.
Groups:
- ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set): On Day 1 (Visit 1), Neisseria meningitidis group A, C, W, and Y (ACWY) naive participants received a single dose of 0.5 milliliter (mL) Neisseria meningitidis serogroup A, B, C, W, Y (MenABCWY) intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY naive participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of meningococcal (groups A, C, Y, and W-135) oligosaccharide diphtheria conjugate vaccine (MenACWY-CRM) intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3,participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY experienced participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY experienced participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set): On Day 1 (Visit 1), ACWY naive participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2). and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to safety analyses only. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set): On Day 1 (Visit 1), ACWY naive participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to safety analyses only. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set): On Day 1 (Visit 1), ACWY experienced participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to safety analyses only. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set): On Day 1 (Visit 1), ACWY experienced participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to safety analyses only. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
Period: Vaccination Phase (Approx. 7 Months)
Arm/Group | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set) | ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set) | ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set) | ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set)
Started | 552 | 276 | 528 | 261 (One participant initially randomized to group 3 was included in group 4 as participant received the wrong vaccination (Trumenba + saline).) | 544 | 57 | 154 | 59
Vaccination 1 | 547 | 274 | 526 | 261 | 537 | 56 | 153 | 59
Vaccination 2 | 500 | 254 | 453 | 218 | 481 | 46 | 123 | 45
Completed | 490 | 248 | 440 | 209 | 476 | 45 | 122 | 44
Not Completed | 62 | 28 | 88 | 52 | 68 | 12 | 32 | 15
Not completed — Lost to Follow-up | 26 | 15 | 42 | 22 | 30 | 3 | 18 | 5
Not completed — Medication error without associated adverse event | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 5 | 1 | 5 | 2 | 3 | 0 | 2 | 3
Not completed — Pregnancy | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 5 | 3 | 0 | 0 | 3 | 0
Not completed — Other | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 18 | 14 | 10 | 3 | 5 | 4
Not completed — Withdrawal by parent/guardian | 10 | 4 | 11 | 7 | 16 | 4 | 3 | 2
Not completed — Withdrawn before vaccination | 5 | 2 | 2 | 0 | 7 | 1 | 1 | 0
Period: Follow-up Phase (Approx. 5 Months)
Arm/Group | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set) | ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set) | ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set) | ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set)
Started | 490 | 248 | 440 | 209 | 476 | 45 | 122 | 44
Completed | 487 | 243 | 440 | 208 | 475 | 45 | 120 | 43
Not Completed | 3 | 5 | 0 | 1 | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 3 | 5 | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination. One participant initially randomized to group 3 was excluded from safety population set as the participant received the wrong vaccination (Trumenba + saline).
Groups:
- ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY naive participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY naive participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY experienced participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. . Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set): On Day 1 (Visit 1), ACWY naive participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to safety analyses only. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- Total: Total of all reporting groups
Arm/Group | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set) | ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set) | ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set) | ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set) | Total
Number analyzed (Participants) | 547 | 274 | 526 | 260 | 537 | 56 | 153 | 59 | 2412
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.7 (5.49) | 16.7 (5.39) | 17.3 (3.17) | 17.4 (3.28) | 13.5 (4.05) | 13.5 (4.50) | 17.1 (3.04) | 16.0 (2.75) | 16.1 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289 | 140 | 279 | 131 | 253 | 20 | 96 | 28 | 1236
  Male | 258 | 134 | 247 | 129 | 284 | 36 | 57 | 31 | 1176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 53 | 156 | 86 | 131 | 15 | 58 | 29 | 621
  Not Hispanic or Latino | 450 | 217 | 366 | 173 | 405 | 41 | 93 | 30 | 1775
  Unknown or Not Reported | 4 | 4 | 4 | 1 | 1 | 0 | 2 | 0 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 2 | 4 | 1 | 2 | 1 | 16
  Asian | 19 | 4 | 18 | 6 | 7 | 1 | 1 | 1 | 57
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 4
  Black or African American | 26 | 19 | 74 | 32 | 57 | 5 | 27 | 5 | 245
  White | 467 | 239 | 370 | 195 | 419 | 46 | 103 | 42 | 1881
  More than one race | 9 | 3 | 12 | 3 | 7 | 2 | 2 | 0 | 38
  Unknown or Not Reported | 23 | 7 | 48 | 22 | 42 | 1 | 18 | 10 | 171

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving At Least 4-Fold Rise in Serum Bactericidal Assay Using Human Complement (hSBA) Titer From Baseline for Each MenACWY Strains: 1 Month After Vaccination 2 in Group 1 Compared to 1 Month After Vaccination 1 in Group 2
Description: 4-fold increase was defined as: 1) for participants with baseline hSBA titer below limit of detection (LOD) (or hSBA titer less than [<] 1:4), 4-fold rise was defined as hSBA titer greater than or equal to (>=) 1:16; 2) baseline hSBA titer >=LOD and < lower limit of quantitation (LLOQ) (i.e. hSBA titer of 1:8), 4-fold rise was defined as hSBA titer >=4 times LLOQ; 3) baseline hSBA titer >=LLOQ, 4-fold rise was defined as hSBA titer >=4 times baseline titer. Exact 2-sided confidence interval (CI) using Clopper and Pearson method was presented. Analysis was performed on post-vaccination (PV) 1 evaluable immunogenicity population (EIP) for Group 2 and PV2 evaluable immunogenicity population for Group 1. Here, 'Overall Number of Participants Analyzed' represented as 'N' and 'Number Analyzed' represented as 'n'.
Time Frame: Baseline (pre-vaccination on Day 1), 1 month after Vaccination 2 in Group 1 and 1 month after Vaccination 1 in Group 2
Population: PV1 EIP and PV2 EIP: randomized to study group of interest; eligible at visit (V) 2 and 4 respectively; received vaccine at V1 or V1 and V3, respectively; blood drawn for assay testing at specified time points; at least 1 valid, determinate MenACWY or MenACWY/MenB assay result; no prohibited vaccine/treatment, no protocol deviations through V2 and V4, respectively. N=participants evaluable for outcome measure; n=participants evaluable for rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set)
Number analyzed (Participants) | 451 | 254
Percentage of participants
  MenA: number analyzed (Participants) | 447 | 254
  MenA | 97.8 [95.9 to 98.9] | 95.3 [91.9 to 97.5]
  MenC: number analyzed (Participants) | 451 | 252
  MenC | 93.3 [90.6 to 95.5] | 52.4 [46.0 to 58.7]
  MenW: number analyzed (Participants) | 439 | 244
  MenW | 97.3 [95.3 to 98.6] | 73.0 [66.9 to 78.4]
  MenY: number analyzed (Participants) | 446 | 248
  MenY | 94.4 [91.8 to 96.3] | 70.6 [64.5 to 76.2]
Statistical Analysis 1: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenA; Test type: Non-Inferiority — 95% CI for the difference in percentage of participants was calculated based on Miettinen and Nurminen. If the lower limit of the 2-sided 95% CI for the difference in percentage of participants was greater than (>) minus (-)10 percent (%), the non-inferiority was concluded; Based on Miettinen and Nurminen method; Difference in percentage of participants = 2.5, 95% CI 2-sided [-0.2 to 6.0]
Statistical Analysis 2: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenC; Test type: Non-Inferiority — 95% CI for the difference in percentage of participants was calculated based on Miettinen and Nurminen. If the lower limit of the 2-sided 95% CI for the difference in percentage of participants was > -10%, the non-inferiority was concluded; Difference in percentage of participants = 41.0, 95% CI 2-sided [34.4 to 47.5]
Statistical Analysis 3: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenW; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 24.3, 95% CI 2-sided [18.8 to 30.4]
Statistical Analysis 4: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenY; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 23.8, 95% CI 2-sided [18.0 to 30.1]

2. Primary Outcome: Percentage of Participants Achieving At Least 4-Fold Rise in hSBA Titer From Baseline for Each of the MenACWY Strains: 1 Month After Vaccination 2 in Group 3 Compared to 1 Month After Vaccination 1 in Group 4
Description: 4-fold increase was defined as: 1) for participants with baseline hSBA titer below LOD (or hSBA titer <1:4), 4-fold rise was defined as hSBA titer >=1:16; 2) baseline hSBA titer >=LOD (i.e., hSBA titer of >=1:4) and < LLOQ (i.e., hSBA titer of 1:8), 4-fold rise was defined as hSBA titer >=4times LLOQ; 3) baseline hSBA titer >=LLOQ, 4-fold rise was defined as hSBA titer >=4 times baseline titer. Exact 2-sided CI using Clopper and Pearson method was presented. Here, 'Overall Number of Participants Analyzed' represented as 'N' and 'Number Analyzed' represented as 'n'.
Time Frame: Baseline (pre-vaccination on Day 1), 1 month after Vaccination 2 in Group 3 and 1 month after Vaccination 1 in Group 4
Population: PV1 and PV2 EIP for Group 4 and Group 3, respectively: randomized to study group of interest; eligible at V2 and V4, respectively; received vaccine at V1 or V1 and V3, respectively; blood drawn for assay testing at specified time points; at least 1 valid, determinate MenACWY or MenACWY/MenB assay result, no prohibited vaccines/treatment, no protocol deviations through V2 and V4 respectively. N=participants evaluable for outcome measure; n=participants evaluable for rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set)
Number analyzed (Participants) | 387 | 227
Percentage of participants
  MenA: number analyzed (Participants) | 385 | 227
  MenA | 93.8 [90.9 to 96.0] | 96.9 [93.7 to 98.8]
  MenC: number analyzed (Participants) | 386 | 226
  MenC | 93.8 [90.9 to 96.0] | 94.7 [90.9 to 97.2]
  MenW: number analyzed (Participants) | 386 | 222
  MenW | 97.1 [94.8 to 98.5] | 96.4 [93.0 to 98.4]
  MenY: number analyzed (Participants) | 387 | 223
  MenY | 93.0 [90.0 to 95.4] | 93.7 [89.7 to 96.5]
Statistical Analysis 1: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenA; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = -3.2, 95% CI 2-sided [-6.5 to 0.5]
Statistical Analysis 2: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenC; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = -0.9, 95% CI 2-sided [-4.6 to 3.3]
Statistical Analysis 3: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenW; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 0.7, 95% CI 2-sided [-2.2 to 4.3]
Statistical Analysis 4: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenY; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = -0.7, 95% CI 2-sided [-4.6 to 3.8]

3. Primary Outcome: Percentage of Participants Achieving hSBA Titer Greater Than or Equal to (>=) LLOQ for All Primary Neisseria Meningitidis Group B (MenB) Test Strains Combined (Composite Response): Groups 1 and 3 Combined Versus Groups 2 and 4 Combined
Description: Percentage of participants achieving hSBA titer >= LLOQ (1:16 for strain A22 and 1:8 for strains A56, B24, and B44) for all MenB test strains (A22, A56, B24 and B44) combined were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: 1 month after Vaccination 2
Population: PV2 EIP: participants randomized to study group of interest; eligible at V4; received vaccine at V1 and V3; blood drawn for assay testing at specified time points; had at least 1 valid, determinate MenACWY or MenB assay result at V4; received no prohibited vaccines; no protocol deviations through V4. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY naive and ACWY experienced participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set): On Day 1 (Visit 1), ACWY naive and ACWY experienced participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination and contributed to both safety and immunogenicity analyses. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
Arm/Group | Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) | Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set)
Number analyzed (Participants) | 755 | 383
Percentage of participants | 78.3 [75.2 to 81.2] | 68.7 [63.8 to 73.3]
Statistical Analysis 1: Comparison: Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) vs Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 9.6, 95% CI 2-sided [4.2 to 15.2]

4. Primary Outcome: Percentage of Participants Achieving At Least a 4-Fold Rise in hSBA Titer From Baseline For Each Primary MenB Test Strains at 1 Month After Vaccination 2: Groups 1 and 3 Combined Versus Groups 2 and 4 Combined
Description: Percentage of participants achieving at least a 4-fold rise in hSBA titer for each primary MenB test strains (A22, A56, B24 and B44) were reported in this outcome measure. Exact 2-sided CI using the Clopper and Pearson method was presented.
Time Frame: Baseline (pre-vaccination on Day 1), 1 month after Vaccination 2
Population: PV2 EIP: participants randomized to study group of interest; eligible at V4; received vaccine at V1 and V3; blood drawn for assay testing at specified time points; at least 1 valid, determinate MenACWY or MenB assay result at V4; no prohibited vaccines; no protocol deviations through V4. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for outcome measure and 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) | Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set)
Number analyzed (Participants) | 845 | 419
Percentage of participants
  A22: number analyzed (Participants) | 778 | 396
  A22 | 83.0 [80.2 to 85.6] | 79.0 [74.7 to 82.9]
  A56: number analyzed (Participants) | 807 | 400
  A56 | 95.9 [94.3 to 97.2] | 94.5 [91.8 to 96.5]
  B24: number analyzed (Participants) | 833 | 418
  B24 | 68.1 [64.8 to 71.2] | 57.2 [52.3 to 62.0]
  B44 | 86.5 [84.0 to 88.7] | 79.2 [75.0 to 83.0]
Statistical Analysis 1: Comparison: Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) vs Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set); A22; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 4.0, 95% CI 2-sided [-0.7 to 8.9]
Statistical Analysis 2: Comparison: Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) vs Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set); A56; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 1.4, 95% CI 2-sided [-1.0 to 4.3]
Statistical Analysis 3: Comparison: Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) vs Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set); B24; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 10.9, 95% CI 2-sided [5.2 to 16.6]
Statistical Analysis 4: Comparison: Groups 1+3 Combined MenABCWY + Saline (Immunogenicity and Safety Set) vs Groups 2+4 Combined Trumenba + MenACWY-CRM (Immunogenicity and Safety Set); B44; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 7.3, 95% CI 2-sided [2.9 to 11.9]

5. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units. 1 caliper unit =0.5 centimeter (cm) and graded as mild: >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity. Percentage of participants with local reactions at injection site were reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after Vaccination 1
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination. Here, "Overall Number of Participants Analyzed" (N) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Groups 1+3+5+7 Combined MenABCWY + Saline: On Day 1 (Visit 1), ACWY naive and ACWY experienced participants received a single dose of 0.5 mL MenABCWY intramuscularly into the left deltoid muscle along with 0.5 mL of saline intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of MenABCWY intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
- Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM: On Day 1 (Visit 1), ACWY naive and ACWY experienced participants received a single dose of 0.5 mL Trumenba intramuscularly into the left deltoid muscle along with 0.5 mL of MenACWY-CRM intramuscularly into the right deltoid muscle (Vaccination 1). Participants were followed up for 1 month after Vaccination 1 (Visit 2). After 6 months of Vaccination 1 at Visit 3, participants received 0.5 mL of Trumenba intramuscularly into the left deltoid muscle (Vaccination 2) and were followed up for 1 month after Vaccination 2 (Visit 4). Vaccination phase was from Day 1 of Vaccination 1 through 1 month after Vaccination 2 (from Visit 1 to Visit 4). Participants were followed up for 6 months after last vaccination. Follow-up phase was from 1 month after Vaccination 2 through 6 months after Vaccination 2.
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1722 | 630
Percentage of participants
  Redness: Mild | 8.8 [7.5 to 10.3] | 7.3 [5.4 to 9.6]
  Redness: Moderate | 14.5 [12.8 to 16.2] | 10.0 [7.8 to 12.6]
  Redness: Severe | 2.5 [1.8 to 3.3] | 2.2 [1.2 to 3.7]
  Swelling: Mild | 10.5 [9.0 to 12.0] | 8.3 [6.2 to 10.7]
  Swelling: Moderate | 13.3 [11.7 to 15.0] | 12.4 [9.9 to 15.2]
  Swelling: Severe | 1.2 [0.7 to 1.8] | 0.8 [0.3 to 1.8]
  Pain at injection site: Mild | 32.3 [30.1 to 34.6] | 31.1 [27.5 to 34.9]
  Pain at injection site: Moderate | 49.5 [47.1 to 51.9] | 47.6 [43.7 to 51.6]
  Pain at injection site: Severe | 7.5 [6.3 to 8.8] | 6.3 [4.6 to 8.5]

6. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an e-diary. Redness and swelling were measured and recorded in caliper units. 1 caliper unit =0.5 cm and graded as mild: >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity. Percentage of participants with local reactions at injection site were reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after Vaccination 2
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1456 | 529
Percentage of participants
  Redness: Mild | 7.7 [6.4 to 9.2] | 6.6 [4.7 to 9.1]
  Redness: Moderate | 12.6 [10.9 to 14.4] | 7.2 [5.1 to 9.7]
  Redness: Severe | 3.0 [2.1 to 4.0] | 0.9 [0.3 to 2.2]
  Swelling: Mild | 10.4 [8.9 to 12.1] | 6.4 [4.5 to 8.9]
  Swelling: Moderate | 12.8 [11.1 to 14.6] | 8.1 [5.9 to 10.8]
  Swelling: Severe | 1.0 [0.5 to 1.6] | 0.2 [0.0 to 1.0]
  Pain at injection site: Mild | 29.1 [26.7 to 31.5] | 33.1 [29.1 to 37.3]
  Pain at injection site: Moderate | 48.8 [46.2 to 51.4] | 40.3 [36.1 to 44.6]
  Pain at injection site: Severe | 6.5 [5.3 to 7.9] | 5.3 [3.5 to 7.6]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: Systemic events were recorded by participants in e-diary. Fever was defined as temperature >=38.0 degrees (deg) Celsius (C) and was categorized as 38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after Vaccination 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1739 | 638
Percentage of participants
  Fever: 38.0 deg C to 38.4 deg C | 3.7 [2.8 to 4.7] | 2.0 [1.1 to 3.5]
  Fever: >38.4 deg C to 38.9 deg C | 1.6 [1.0 to 2.3] | 2.8 [1.7 to 4.4]
  Fever: >38.9 deg C to 40.0 deg C | 0.6 [0.3 to 1.1] | 0.9 [0.3 to 2.0]
  Fever: >40.0 deg C | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.6]
  Fatigue: Mild | 23.5 [21.5 to 25.5] | 25.7 [22.4 to 29.3]
  Fatigue: Moderate | 25.5 [23.4 to 27.6] | 25.7 [22.4 to 29.3]
  Fatigue: Severe | 3.2 [2.4 to 4.1] | 3.3 [2.0 to 5.0]
  Headache: Mild | 25.6 [23.6 to 27.8] | 24.5 [21.2 to 28.0]
  Headache: Moderate | 19.2 [17.4 to 21.1] | 20.4 [17.3 to 23.7]
  Headache: Severe | 1.9 [1.3 to 2.7] | 2.0 [1.1 to 3.5]
  Chills: Mild | 12.6 [11.1 to 14.2] | 10.2 [8.0 to 12.8]
  Chills: Moderate | 6.7 [5.5 to 7.9] | 7.8 [5.9 to 10.2]
  Chills: Severe | 0.8 [0.4 to 1.3] | 1.6 [0.8 to 2.9]
  Vomiting: Mild | 2.5 [1.8 to 3.4] | 2.0 [1.1 to 3.5]
  Vomiting: Moderate | 0.6 [0.3 to 1.1] | 0.9 [0.3 to 2.0]
  Vomiting: Severe | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.6]
  Diarrhea: Mild | 8.7 [7.5 to 10.2] | 11.9 [9.5 to 14.7]
  Diarrhea: Moderate | 2.0 [1.4 to 2.7] | 1.6 [0.8 to 2.9]
  Diarrhea: Severe | 0.3 [0.1 to 0.7] | 0.0 [0.0 to 0.6]
  Muscle Pain: Mild | 13.6 [12.0 to 15.3] | 13.5 [10.9 to 16.4]
  Muscle Pain: Moderate | 10.5 [9.1 to 12.1] | 11.9 [9.5 to 14.7]
  Muscle Pain: Severe | 1.6 [1.1 to 2.3] | 2.0 [1.1 to 3.5]
  Joint Pain: Mild | 10.7 [9.3 to 12.2] | 12.9 [10.4 to 15.7]
  Joint Pain: Moderate | 8.6 [7.3 to 10.0] | 8.6 [6.6 to 11.1]
  Joint Pain: Severe | 1.0 [0.6 to 1.6] | 1.1 [0.4 to 2.2]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: Systemic events were recorded by participants in e-diary. Fever was defined as temperature >=38.0 deg C and was categorized as 38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24h, moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1459 | 532
Percentage of participants
  Fever: 38.0 deg C to 38.4 deg C | 1.8 [1.2 to 2.6] | 0.4 [0.0 to 1.4]
  Fever: >38.4 deg C to 38.9 deg C | 0.3 [0.1 to 0.7] | 0.9 [0.3 to 2.2]
  Fever: >38.9 deg C to 40.0 deg C | 0.2 [0.0 to 0.6] | 0.2 [0.0 to 1.0]
  Fever: >40.0 deg C | 0.0 [0.0 to 0.3] | 0.0 [0.0 to 0.7]
  Fatigue: Mild | 22.8 [20.7 to 25.1] | 22.0 [18.5 to 25.8]
  Fatigue: Moderate | 21.8 [19.7 to 24.0] | 19.9 [16.6 to 23.6]
  Fatigue: Severe | 2.9 [2.1 to 3.9] | 1.7 [0.8 to 3.2]
  Headache: Mild | 21.3 [19.2 to 23.5] | 21.1 [17.7 to 24.8]
  Headache: Moderate | 16.8 [14.9 to 18.8] | 16.2 [13.1 to 19.6]
  Headache: Severe | 1.7 [1.1 to 2.5] | 0.6 [0.1 to 1.6]
  Chills: Mild | 9.9 [8.5 to 11.6] | 8.8 [6.6 to 11.6]
  Chills: Moderate | 6.0 [4.9 to 7.4] | 5.8 [4.0 to 8.2]
  Chills: Severe | 0.4 [0.2 to 0.9] | 1.5 [0.7 to 2.9]
  Vomiting: Mild | 1.4 [0.8 to 2.1] | 0.8 [0.2 to 1.9]
  Vomiting: Moderate | 0.1 [0.0 to 0.5] | 0.2 [0.0 to 1.0]
  Vomiting: Severe | 0.0 [0.0 to 0.3] | 0.0 [0.0 to 0.7]
  Diarrhea: Mild | 6.9 [5.6 to 8.3] | 6.0 [4.2 to 8.4]
  Diarrhea: Moderate | 1.4 [0.8 to 2.1] | 2.4 [1.3 to 4.1]
  Diarrhea: Severe | 0.0 [0.0 to 0.3] | 0.0 [0.0 to 0.7]
  Muscle Pain: Mild | 10.0 [8.5 to 11.7] | 10.0 [7.6 to 12.8]
  Muscle Pain: Moderate | 11.9 [10.3 to 13.7] | 11.5 [8.9 to 14.5]
  Muscle Pain: Severe | 0.8 [0.4 to 1.4] | 0.8 [0.2 to 1.9]
  Joint Pain: Mild | 9.6 [8.1 to 11.2] | 7.9 [5.7 to 10.5]
  Joint Pain: Moderate | 8.3 [6.9 to 9.8] | 6.8 [4.8 to 9.2]
  Joint Pain: Severe | 0.4 [0.2 to 0.9] | 0.9 [0.3 to 2.2]

9. Primary Outcome: Percentage of Participants With Use of Antipyretic Medication Within 7 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: The use of antipyretic medication was recorded by participants in an e-diary for 7 days after vaccination. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after Vaccination 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1739 | 638
Percentage of participants | 29.5 [27.4 to 31.7] | 28.1 [24.6 to 31.7]

10. Primary Outcome: Percentage of Participants With Use of Antipyretic Medication Within 7 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: The use of antipyretic medication recorded by participants in an e-diary for 7 days after vaccination. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1459 | 532
Percentage of participants | 25.1 [22.9 to 27.4] | 20.5 [17.1 to 24.2]

11. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 30 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. Exact 2-sided CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Within 30 days after Vaccination 1
Population: Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 5.8 [4.7 to 7.0] | 6.5 [4.7 to 8.6]

12. Primary Outcome: Percentage of Participants With AEs Within 30 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 11
Time Frame: Within 30 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1558 | 562
Percentage of participants | 5.3 [4.3 to 6.6] | 3.7 [2.3 to 5.7]

13. Primary Outcome: Percentage of Participants With AEs Within 30 Days After Any Vaccination: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 11
Time Frame: Within 30 days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 9.7 [8.4 to 11.2] | 9.1 [7.0 to 11.6]

14. Primary Outcome: Percentage of Participants With AEs During Vaccination Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 11
Time Frame: From day of Vaccination 1 (Day 1) up to 1 month after Vaccination 2 (approximately 7 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 20.9 [19.0 to 22.8] | 20.3 [17.3 to 23.6]

15. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 30 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/incapacity; congenital anomaly/birth defect and other important medical events. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after Vaccination 1
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0.06 [0.0 to 0.3] | 0.0 [0.0 to 0.6]

16. Primary Outcome: Percentage of Participants With SAEs Within 30 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 15
Time Frame: Within 30 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1558 | 562
Percentage of participants | 0.1 [0.0 to 0.5] | 0.0 [0.0 to 0.7]

17. Primary Outcome: Percentage of Participants With SAEs Within 30 Days After Any Vaccination: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent disability/ incapacity; congenital anomaly/birth defect and other important medical events. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0.2 [0.0 to 0.5] | 0.0 [0.0 to 0.6]

18. Primary Outcome: Percentage of Participants With SAEs During Vaccination Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 17
Time Frame: From day of Vaccination 1 (Day 1) up to 1 month after Vaccination 2 (approximately 7 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0.4 [0.2 to 0.8] | 0.0 [0.0 to 0.6]

19. Primary Outcome: Percentage of Participants With SAEs During Follow-up Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 17
Time Frame: From 1 month after Vaccination 2 up to 6 months after Vaccination 2 (approximately 5 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1390 | 509
Percentage of participants | 0.3 [0.1 to 0.7] | 0.8 [0.2 to 2.0]

20. Primary Outcome: Percentage of Participants With SAEs Throughout the Study: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 17
Time Frame: From day of Vaccination 1 (Day 1) up to 6 months after Vaccination 2 (approximately 12 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0.6 [0.3 to 1.1] | 0.6 [0.2 to 1.6]

21. Primary Outcome: Percentage of Participants With Medically Attended Adverse Events (MAEs) Within 30 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after Vaccination 1
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 3.6 [2.8 to 4.5] | 4.3 [2.9 to 6.2]

22. Primary Outcome: Percentage of Participants With MAEs Within 30 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 21
Time Frame: Within 30 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1558 | 562
Percentage of participants | 3.6 [2.7 to 4.6] | 2.8 [1.6 to 4.6]

23. Primary Outcome: Percentage of Participants With MAEs Within 30 Days After Any Vaccination: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 21
Time Frame: Within 30 days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 6.3 [5.2 to 7.5] | 6.3 [4.6 to 8.5]

24. Primary Outcome: Percentage of Participants With MAEs During Vaccination Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 21
Time Frame: From day of Vaccination 1 (Day 1) up to 1 month after Vaccination 2 (approximately 7 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 14.9 [13.3 to 16.7] | 14.3 [11.7 to 17.3]

25. Primary Outcome: Percentage of Participants With MAEs During Follow-up Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 21
Time Frame: From 1 month after Vaccination 2 up to 6 months after Vaccination 2 (approximately 5 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1390 | 509
Percentage of participants | 9.3 [7.8 to 10.9] | 7.5 [5.3 to 10.1]

26. Primary Outcome: Percentage of Participants With MAEs Throughout the Study: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 21
Time Frame: From day of Vaccination 1 (Day 1) up to 6 months after Vaccination 2 (approximately 12 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 19.3 [17.5 to 21.2] | 18.3 [15.4 to 21.5]

27. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition (NDCMC) Within 30 Days After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 days after Vaccination 1
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0.2 [0.1 to 0.6] | 0.0 [0.0 to 0.6]

28. Primary Outcome: Percentage of Participants With NDCMC Within 30 Days After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 27
Time Frame: Within 30 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1558 | 562
Percentage of participants | 0.06 [0.0 to 0.4] | 0.0 [0.0 to 0.7]

29. Primary Outcome: Percentage of Participants With NDCMC Within 30 Days After Any Vaccination: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 27
Time Frame: Within 30 Days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0.3 [0.1 to 0.7] | 0.0 [0.0 to 0.6]

30. Primary Outcome: Percentage of Participants With NDCMC During Vaccination Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 27
Time Frame: From day of Vaccination 1 (Day 1) up to 1 month after Vaccination 2 (approximately 7 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 1.1 [0.7 to 1.7] | 0.3 [0.0 to 1.1]

31. Primary Outcome: Percentage of Participants With NDCMC During Follow-up Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 27
Time Frame: From 1 month after Vaccination 2 up to 6 months after Vaccination 2 (approximately 5 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1390 | 509
Percentage of participants | 0.4 [0.1 to 0.8] | 0.0 [0.0 to 0.7]

32. Primary Outcome: Percentage of Participants With NDCMC Throughout the Study: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 27
Time Frame: From day of Vaccination 1 (Day 1) up to 6 months after Vaccination 2 (approximately 12 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 1.4 [0.9 to 2.1] | 0.3 [0.0 to 1.1]

33. Primary Outcome: Percentage of Participants With Immediate AE Within 30 Minutes After Vaccination 1: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: Immediate AEs were defined as AEs occurring within the first 30 minutes after investigational product administration. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Within 30 minutes after Vaccination 1
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 0 [NA to NA] — Lower and upper limit of 95% CI could not be estimated, due to insufficient participants with event. | 0 [NA to NA] — Lower and upper limit of 95% CI could not be estimated, due to insufficient participants with event.

34. Primary Outcome: Percentage of Participants With Immediate AE Within 30 Minutes After Vaccination 2: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: as for outcome 33
Time Frame: Within 30 minutes after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1558 | 562
Percentage of participants | 0 [NA to NA] — Lower and upper limit of 95% CI could not be estimated, due to insufficient participants with event. | 0 [NA to NA] — Lower and upper limit of 95% CI could not be estimated, due to insufficient participants with event.

35. Primary Outcome: Percentage of Participants Who Missed Days of School or Work Due to AEs During Vaccination Phase: By MenABCWY Group (Groups 1, 3, 5, and 7 Combined) and Trumenba Group (Groups 2, 4, 6, and 8 Combined)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of investigational product, whether or not considered related to the investigational product. Percentage of participants who missed days of school or work due to AEs during vaccination phase were reported in this outcome measure.
Time Frame: From day of Vaccination 1 (Day 1) up to 1 month after Vaccination 2 (approximately 7 months)
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Groups 1+3+5+7 Combined MenABCWY + Saline | Groups 2+4+6+8 Combined Trumenba + MenACWY-CRM
Number analyzed (Participants) | 1763 | 649
Percentage of participants | 5.0 | 4.5

36. Secondary Outcome: Percentage of Participants Achieving At Least 4-Fold Rise in hSBA Titer From Baseline for Each MenACWY Test Strains: 1 Month After Vaccination 1 in Group 1 Compared to Group 2
Description: 4-fold increase was defined as: 1) for participants with baseline hSBA titer below LOD (or hSBA titer <1:4), 4-fold rise was defined as hSBA titer >=1:16; 2) baseline hSBA titer >=LOD (i.e., hSBA titer of >=1:4) and < LLOQ (i.e. hSBA titer of 1:8), 4-fold rise was defined as hSBA titer >=4times LLOQ; 3) baseline hSBA titer >=LLOQ, 4-fold rise was defined as hSBA titer >=4 times baseline titer. Exact 2-sided CI using Clopper and Pearson method was presented.
Time Frame: Baseline (pre-vaccination on Day 1), 1 month after Vaccination 1
Population: PV1 EIP: participants randomized to study group of interest; eligible at V2; received vaccine at V1; blood drawn for assay testing at specified time points; at least 1 valid, determinate MenACWY assay result at V2; no prohibited vaccines; no protocol deviations through V2. Here "Overall Number of Participants Analyzed" = participants evaluable for outcome measure and "Number Analyzed" = number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set)
Number analyzed (Participants) | 501 | 254
Percentage of participants
  MenA: number analyzed (Participants) | 499 | 254
  MenA | 97.0 [95.1 to 98.3] | 95.3 [91.9 to 97.5]
  MenC: number analyzed (Participants) | 501 | 252
  MenC | 62.9 [58.5 to 67.1] | 52.4 [46.0 to 58.7]
  MenW: number analyzed (Participants) | 492 | 244
  MenW | 79.3 [75.4 to 82.8] | 73.0 [66.9 to 78.4]
  MenY: number analyzed (Participants) | 494 | 248
  MenY | 82.0 [78.3 to 85.3] | 70.6 [64.5 to 76.2]
Statistical Analysis 1: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenA; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 1.7, 95% CI 2-sided [-1.0 to 5.3]
Statistical Analysis 2: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenC; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 10.5, 95% CI 2-sided [3.0 to 17.9]
Statistical Analysis 3: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenW; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 6.3, 95% CI 2-sided [-0.1 to 13.1]
Statistical Analysis 4: Comparison: ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenY; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 11.4, 95% CI 2-sided [5.0 to 18.2]

37. Secondary Outcome: Percentage of Participants Achieving At Least 4-Fold Rise in hSBA Titer From Baseline for Each MenACWY Test Strains: 1 Month After Vaccination 1 in Group 3 Compared to Group 4
Description: 4-fold increase was defined as: 1) for participants with baseline hSBA titer below LOD (or hSBA titer <1:4), 4-fold rise was defined as hSBA titer >=1:16; 2) baseline hSBA titer >=LOD (i.e., hSBA titer of >=1:4) and < LLOQ (i.e. hSBA titer of 1:8), 4-fold rise was defined as hSBA titer >=4 times LLOQ; 3) baseline hSBA titer > =LLOQ, 4-fold rise was defined as hSBA titer >=4 times baseline titer. Exact 2-sided CI using Clopper and Pearson method was presented.
Time Frame: Baseline (pre-vaccination on Day 1), 1 month after Vaccination 1
Population: PV1 EIP: participants randomised to study group of interest; eligible at V 2; received vaccine at V1; blood drawn for assay testing at specified time points; at least 1 valid, determinate MenACWY assay result at V2; no prohibited vaccines and no protocol deviations through V2. Here "Overall Number of Participants Analyzed" = participants evaluable for outcome measure and "Number Analyzed" = number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set)
Number analyzed (Participants) | 442 | 227
Percentage of participants
  MenA: number analyzed (Participants) | 439 | 227
  MenA | 94.8 [92.2 to 96.7] | 96.9 [93.7 to 98.8]
  MenC: number analyzed (Participants) | 439 | 226
  MenC | 93.4 [90.7 to 95.5] | 94.7 [90.9 to 97.2]
  MenW: number analyzed (Participants) | 428 | 222
  MenW | 97.4 [95.4 to 98.7] | 96.4 [93.0 to 98.4]
  MenY: number analyzed (Participants) | 442 | 223
  MenY | 94.3 [91.8 to 96.3] | 93.7 [89.7 to 96.5]
Statistical Analysis 1: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenA; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = -2.2, 95% CI 2-sided [-5.2 to 1.4]
Statistical Analysis 2: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenC; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = -1.3, 95% CI 2-sided [-4.9 to 2.9]
Statistical Analysis 3: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenW; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 1.0, 95% CI 2-sided [-1.6 to 4.6]
Statistical Analysis 4: Comparison: ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) vs ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set); MenY; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage of participants = 0.6, 95% CI 2-sided [-3.0 to 5.0]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events recorded using systematic assessment within 7 days after Vaccination 1 and 2; SAEs and all-cause mortality recorded using non-systematic assessment from Day 1 up to 6 months after vaccination 2 (approximately 12 months) and other AEs recorded using non-systematic assessment from Day 1 up to 1 month after vaccination 2 (approximately 7 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population included all randomized participants who received at least 1 dose of investigational product and had safety data reported after vaccination.
Arm/Group | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) | ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set) | ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set) | ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set) | ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set)
All-Cause Mortality (participants affected / at risk) | 0/547 | 0/274 | 0/526 | 0/260 | 0/537 | 0/56 | 0/153 | 0/59
Serious Adverse Events (participants affected / at risk) | 6/547 | 1/274 | 3/526 | 2/260 | 2/537 | 1/56 | 0/153 | 0/59
Other Adverse Events (participants affected / at risk) | 533/547 | 262/274 | 504/526 | 244/260 | 512/537 | 53/56 | 148/153 | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) (N=547) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) (N=274) | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) (N=526) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) (N=260) | ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set) (N=537) | ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set) (N=56) | ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set) (N=153) | ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set) (N=59)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Status migrainosus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACWY-Naive: Group 1 MenABCWY + Saline (Immunogenicity and Safety Set) (N=547) | ACWY-Naive: Group 2 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) (N=274) | ACWY-Experienced: Group 3 MenABCWY + Saline (Immunogenicity and Safety Set) (N=526) | ACWY-Experienced: Group 4 Trumenba+ MenACWY - CRM (Immunogenicity and Safety Set) (N=260) | ACWY-Naive: Group 5 MenABCWY + Saline (Safety Set) (N=537) | ACWY-Naive: Group 6 Trumenba+ MenACWY - CRM (Safety Set) (N=56) | ACWY-Experienced: Group 7 MenABCWY + Saline (Safety Set) (N=153) | ACWY-Experienced: Group 8 Trumenba+ MenACWY - CRM (Safety Set) (N=59)
Cerumen impaction (Ear and labyrinth disorders) | 2 | 1 | 4 | 2 | 2 | 0 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 5 | 1 | 2 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 6 | 0 | 3 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 69 | 50 | 116 | 54 | 72 | 8 | 23 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Vomiting (VOMITING) (Gastrointestinal disorders) | 23 | 13 | 22 | 4 | 21 | 3 | 5 | 3
Chills (CHILLS) (General disorders) | 155 | 78 | 151 | 59 | 130 | 14 | 43 | 19
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Fatigue (FATIGUE) (General disorders) | 364 | 183 | 337 | 160 | 317 | 30 | 99 | 43
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 522 | 247 | 486 | 228 | 493 | 51 | 144 | 57
Pyrexia (General disorders) | 2 | 0 | 2 | 0 | 4 | 0 | 1 | 1
Pyrexia (FEVER) (General disorders) | 44 | 24 | 29 | 13 | 42 | 3 | 8 | 3
Swelling (SWELLING) (General disorders) | 186 | 71 | 158 | 57 | 200 | 16 | 49 | 19
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 22 | 12 | 24 | 12 | 36 | 3 | 10 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 0 | 2 | 0 | 2 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Lice infestation (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 1 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 2 | 4 | 1 | 3 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 5 | 4 | 10 | 2 | 10 | 2 | 7 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 1
Respiratory tract infection viral (Infections and infestations) | 3 | 0 | 1 | 1 | 1 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 5 | 4 | 4 | 0 | 6 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 7 | 17 | 7 | 11 | 4 | 7 | 1
Viral infection (Infections and infestations) | 1 | 2 | 0 | 3 | 3 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1 | 0 | 3 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 6 | 0 | 3 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 2 | 5 | 4 | 6 | 1 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 6 | 0 | 1 | 1 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 4 | 2 | 8 | 3 | 4 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 1 | 1 | 0 | 2 | 2
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 156 | 75 | 156 | 83 | 144 | 12 | 48 | 19
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 198 | 97 | 207 | 97 | 167 | 18 | 57 | 22
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 3 | 3 | 0 | 2 | 1
Headache (HEADACHE) (Nervous system disorders) | 330 | 152 | 312 | 161 | 282 | 24 | 86 | 37
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 0 | 2 | 0 | 2 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 2 | 3 | 0 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 3 | 8 | 0 | 1 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 183 | 75 | 162 | 58 | 190 | 15 | 39 | 16
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT04440163/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT04440163/SAP_001.pdf